CLINICAL TRIAL: NCT03565627
Title: The Feasibility and Acceptability of a Randomised Crossover Trial Assessing Two Current Health Apps for Increasing Physical Activity: a Mixed Methods Study
Brief Title: Feasibility, Acceptability and the Effects of Two Publicly Available Physical Activity Mobile Apps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 11121/001
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: PHYSICAL FITNESS
Keywords: mHealth; digital health; behavior change; physical activity; mobile apps
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will complete a baseline assessment (1 week), followed by the randomisation to using 1 of the 2 apps (3 weeks' follow up), and crossover (5 weeks' follow up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise app (Experimental): 7 Minute Workout Challenge by Fitness Guide Inc.
  Interventions: Device: Exercise app: 7 Minute Workout Challenge
- Running App (Experimental): One You Couch to 5K by Public Health England
  Interventions: Device: Running app: One You Couch to 5K

INTERVENTIONS:
Device: Exercise app: 7 Minute Workout Challenge — 7 Minute Workout Challenge by Fitness Guide Inc. combines aerobic and resistance training into short, 7 minute high intensity circuit training.
  Arms: Exercise app
Device: Running app: One You Couch to 5K — One You Couch to 5K by Public Health England is a popular app that aims to increase fitness by asking the user to follow a running programme with a goal to run for 30 min without break.
  Arms: Running App

SUMMARY:
Within the new digital health care landscape, the rise of health applications (apps) creates novel prospects for behaviour change opportunities. The commercial market is saturated with apps that aim to increase physical activity (PA) with more than 49,000 PA apps available in the major app stores in 2016 [1]. Despite the wide distribution and popularity of PA apps, research on the efficacy of the apps is lacking.

This project focuses on exploring the potential for increasing PA levels using 2 selected apps that are available on the market with participants that do not engage or perform very little PA. This study is timely because PA apps on the market are extremely popular and there is a clear need to this the potential of these potentially convenient, accessible, wide-reaching, and cost-effective technology.

Before a large scale study is conducted, it is crucial to conduct assessment of the feasibility and acceptability of the study [2]. Feasibility determines if the study design, procedures, and the intervention can be executed by the researcher. Acceptability assesses the suitability of the study design, procedures, and the intervention from the perspective of the participants and intervention deliverers [3]. Hence, this mixed-methods feasibility study was designed to inform a decision about whether to proceed to a large-scale study. The aim of this study is to investigate the feasibility and acceptability of a study assessing 2 selected PA apps to inform the design of a definitive RCT, and to assess the effects of the app interventions on PA

DETAILED DESCRIPTION:
The aim of this research project is to investigate the feasibility and acceptability of a study assessing 2 selected PA apps to inform the design of a definitive randomised controlled trial, and to assess the effects of the app interventions on PA.

To address the aim, an explanatory mixed-methods study using quantitative (phase 1) and qualitative (phase 2) design will be used. Target population will be those that do not engage, or engage in low levels, of PA and the investigators will aim at recruiting participants from London and surrounding areas.

The primary objective is to determine the feasibility and acceptability of the trial procedures and the interventions delivered using apps.

The secondary objectives are to explore potential effects of the 2 selected PA apps on behavioural and psychological outcomes, and to assess the usability of the apps.

Phase 1 Phase 1 will utilise a crossover which means that half of the participants will be randomly assigned to use 1 of the 2 apps, while the other half will use the 2nd app. After 2 weeks participants will switch.

Participants will complete a baseline assessment (1 week), followed by the randomisation to using 1 of the 2 apps (2 weeks' follow up), and crossover (4 weeks' follow up). The primary outcome of the study will be average percent increase in activity count and will be measured using accelerometer. The secondary measures include exercise self-efficacy, intentions, apps usability and usage.

Phase 2 Following the end of phase 1, a semi-structured interview will be conducted to explore the acceptability and experiences of using the 2 apps (phase 2). The sample will include participants that took part in the crossover trial and consented to being interviewed. Participants that showed frequent usage of the apps, as well as those who used the app infrequently and/or discontinued using the app will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years' old) identified as "moderately inactive" or "inactive" using General Practice Physical Activity Questionnaire
* as the use of accelerometer requires some maintenance from the researcher, it was necessary to include only users that reside in/around London for practical reasons
* willingness to try the apps assessed in the study (walking and workout app)
* those owning a smartphone, iPhone (operating iOS 6.0 or newer and ) or Android (version 2.3.3 and up

Exclusion Criteria:

* do not speak English
* previous use of the apps of interest
* medical conditions that require special attention when conducting physical activity
* current participation in another research study that targets behaviour change

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-28 (Actual)

PRIMARY OUTCOMES:
Recruitment rates as a percentage of eligible participants that consented to partake in the study | Week 5
  Determined by retention (%)

SECONDARY OUTCOMES:
Retention measured by completeness of data at 5 weeks' follow up | Week 5
  Determined by retention (%)
Acceptability of the trial procedures and the interventions | Week 5
  Semi-structured interviews following the completion of the trial
Change in objectively measured PA from baseline to follow-up | Week 3 and 5
  Measured by hip-worn ActiGraph GT3X+
The difference in PA change between the 2 apps | Week 3 and 5
  Measured by hip-worn ActiGraph GT3X+
Change in self-reported PA | Week 3 and 5
  Using International Physical Activity Questionnaires: short last 7 days self-administered format
Change in exercise self-efficacy | Week 3 and 5
  Measured using Self-Efficacy to Regulate Exercise
Change in PA outcome expectancy measure | Week 3 and 5
  Assessed using Physical Activity Outcome Expectancy Measure
Usability of the apps | Week 3 and 5
  Assessed using System Usability Scale
Change in mood | Week 5
  Assessed daily using PACO app
Usage of apps | Week 13
  Long-term usage of apps will be assessed by asking participants if they have any of the apps on the phones and if they have used it since the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Hamilton, MD, PhD, Principal Investigator — University College, London; Elizabeth Murray, MD, PhD, Study Chair — University College, London
Locations (1):
- eHealth Unit, Research Department of Primary Care and Population Health, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] research2guidance. mHealth app developer economics. The state of the art of mHealth application publishing: research2guidance 2014 [updated 5 May 2016]. Available from: http://research2guidance.com/product/mhealth-app-developer-economics-2014/.
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Feeley N, Cossette S, Cote J, Heon M, Stremler R, Martorella G, Purden M. The importance of piloting an RCT intervention. Can J Nurs Res. 2009 Jun;41(2):85-99. PMID 19650515